CLINICAL TRIAL: NCT04356794
Title: Heart Rate Variability Assessment in Dialysis Patients by Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, Taiwan (Other)
Collaborators: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Jia-Ming Chen, Principal Investigator, China Medical University, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y_105_0300
Record Dates: First submitted 2020-04-10; First posted 2020-04-22 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: RLS
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical electroacupuncture(EA) (Experimental): EA were treated for 4 weeks, 3 times per week.
  Interventions: Other: Acupuncture needle with electrical stimulation
- Sham electroacupuncture (Sham Comparator): Sham acupuncture was performed without stimulation and manipulation to avoid eliciting "De Qi" sensations.It were treated for 4 weeks, 3 times per week.
  Interventions: Other: Sham electroacupuncture

INTERVENTIONS:
Other: Acupuncture needle with electrical stimulation — EA is treated for 4 weeks, 3 times per week.
  Arms: Medical electroacupuncture(EA)
Other: Sham electroacupuncture — Sham EA is treated for 4 weeks, 3 times per week.
  Arms: Sham electroacupuncture

SUMMARY:
Title of the study:Heart Rate Variability Assessment in Dialysis Patients by Acupuncture

Study period: 08/2019 - 07/2021

Institution: the Graduate Institute of Chinese Medical Science, China Medical University/ Changhua Christian Hospital,Taiwan

Aim of the study: To investigate the effect of medical acupuncture in comparison to placebo acupuncture by heart rate variability(HRV)

Design: Prospective randomized trial

Intervention: Experiment group using indwelling fixed needles, N=30 ; Control group using placebo needles, N=30

Outcome measures: International RLS Rating Scale, HRV

DETAILED DESCRIPTION:
RLS occurs in 3-15% of the general population and in 10-30% of patients on maintenance dialysis. End-stage renal disease, a decrease in HRV is typically found, with abnormal HRV being considered an independent risk factor for mortality.While the majority of studies show an initial improvement in symptoms, longer studies and clinical experience show that either treatment efficacy decreases with time, and/or augmentation develops: dopaminergic augmentation has been reported to be the main reason for treatment discontinuation and treatment failure in RLS/WED.

The study randomly assigned to either true acupuncture treatment or placebo/sham acupuncture treatment. Each participant will undergo 12 treatments third-weekly, for a period of 4 weeks. At the end of the eighth treatment session, each participant will again fill out a IRLSRS questionnaire ,ISI and HRV test. At the end of the treatment regimen and 5weeks, participants will again fill out a IRLSRS questionnaire ,ISI and HRV test.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients with RLS
* The symptoms expressed ≧ 3 months and more than twice per week.
* A score of at least 20 corresponding to severe RLS ( International Restless Legs Syndrome Rating Scale, IRLSRS).Dialysis patients with RLS

Exclusion Criteria:

* Idiopathic RLS
* Other movement disorders, various psychiatric and organic disorders, cognitive impairment, or bleeding disorders, on anticoagulant therapy, or cardiac pacemaker.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline International restless legs syndrome rating scale(IRLSRS) at 4 weeks,5weeks | Baseline, 4 weeks, 5weeks
  IRLSRS are scored from 4 for the first (top) answer (usually 'very severe') to 0 for the last answer (usually none). All items are scored. The sum of the item scores serves as the scale score.

SECONDARY OUTCOMES:
Change from Baseline ISI and HRV(LF,HF, RMSSD, PNN50) at 4 weeks, 5weeks | Baseline, 4 weeks, 5weeks
  HRV is the measure of the inconsistent gaps between each heartbeat and is used as an index for different aspects of psychology. HRV is an index of the influence of both the parasympathetic nervous system and the sympathetic nervous systems.

CONTACTS AND LOCATIONS:
Overall Officials: Lun-Chien Lo, PHD, Study Director — China Medical University, Taiwan
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pan W, Wang M, Li M, Wang Q, Kwak S, Jiang W, Yamamoto Y. Actigraph evaluation of acupuncture for treating restless legs syndrome. Evid Based Complement Alternat Med. 2015;2015:343201. doi: 10.1155/2015/343201. Epub 2015 Feb 11. PMID 25763089
- [Background] Cripps MG. Acupuncture for restless legs syndrome in patients previously treated with dopaminergic drugs. Acupunct Med. 2011 Sep;29(3):240-1. doi: 10.1136/acupmed-2011-010039. Epub 2011 Jun 22. No abstract available. PMID 21697212
- [Background] Yildiz A, Yildiz C, Karakurt A. Assessment of cardiac autonomic functions by heart rate variability in patients with restless leg syndrome. Turk Kardiyol Dern Ars. 2018 Apr;46(3):191-196. doi: 10.5543/tkda.2018.33896. PMID 29664425
- [Background] Raissi GR, Forogh B, Ahadi T, Ghahramanpoori S, Ghaboussi P, Sajadi S. Evaluation of Acupuncture in the Treatment of Restless Legs Syndrome: A Randomized Controlled Trial. J Acupunct Meridian Stud. 2017 Oct;10(5):346-350. doi: 10.1016/j.jams.2017.08.004. Epub 2017 Aug 22. PMID 29078970
- [Background] Barone DA, Ebben MR, DeGrazia M, Mortara D, Krieger AC. Heart rate variability in restless legs syndrome and periodic limb movements of Sleep. Sleep Sci. 2017 Apr-Jun;10(2):80-86. doi: 10.5935/1984-0063.20170015. PMID 28966745
- [Background] Cikrikcioglu MA, Hursitoglu M, Erkal H, Kinas BE, Sztajzel J, Cakirca M, Arslan AG, Erek A, Halac G, Tukek T. Oxidative stress and autonomic nervous system functions in restless legs syndrome. Eur J Clin Invest. 2011 Jul;41(7):734-42. doi: 10.1111/j.1365-2362.2010.02461.x. Epub 2011 Jan 20. PMID 21250984
- [Derived] Chen JM, Chiu PF, Chang YJ, Hsu PC, Chang CC, Lo LC. Effect of electroacupuncture on restless legs syndrome (RLS) in hemodialysis patients: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Dec 11;99(50):e23629. doi: 10.1097/MD.0000000000023629. PMID 33327340

DOCUMENTS (2):
  • Study Protocol (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT04356794/Prot_002.pdf
  • Informed Consent Form (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT04356794/ICF_001.pdf